CLINICAL TRIAL: NCT05487664
Title: Determining the Independent and Synergistic Effects of Transcutaneous Auricular Neurostimulation (tAN) on Direct Brain Activation in Healthy Individuals
Brief Title: RM1 Project 2 - tAN fMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00122682
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Auricular Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Auricular Neurostimulation (Active 1) (Active Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -ABVN Only stimulation (15Hz stimulation of cymba conchae)
  Interventions: Device: Transcutaneous Auricular Neruostimulation (tAN)
- Auricular Neurostimulation (Active 2) (Active Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -ATNS Only stimulation (100Hz stimulation of the tragus)
  Interventions: Device: Transcutaneous Auricular Neruostimulation (tAN)
- Auricular Neurostimulation (Active 3) (Active Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Combo stimulation (stimulation of both the 15Hz cymba conchae and 100HZ tragus)
  Interventions: Device: Transcutaneous Auricular Neruostimulation (tAN)
- Auricular Neurostimulation (Sham 1) (Sham Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Sham (15Hz stimulation of the earlobe)
  Interventions: Device: Transcutaneous Auricular Neruostimulation (tAN)
- Auricular Neurostimulation (Sham 2) (Sham Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Sham (100Hz stimulation of the earlobe)
  Interventions: Device: Transcutaneous Auricular Neruostimulation (tAN)

INTERVENTIONS:
Device: Transcutaneous Auricular Neruostimulation (tAN) — The intervention we are studying is called transcutaneous auricular neurostimulation (tAN). tAN is simply electrical nerve stimulation administered at the ear which targets both the auricular branch of the vagus nerve (ABVN) and the auriculotemporal nerve (ATN, a branch of the trigeminal nerve).

SUMMARY:
In this one-visit, randomized, double-blind, sham-controlled trial, we plan to use a novel concurrent transcutaneous auricular neurostimulation (tAN) paradigm during functional magnetic resonance imaging (fMRI) paradigm in 96 individuals to determine whether tAN administered to two cranial nerves simultaneously produces greater neurophysiologic effects than stimulating solely to the auricular branch of the vagus nerve (ABVN) or the auriculotemporal nerve (ATN; branch of trigeminal nerve) alone. Within the MRI scanner, each participant will be connected to a series of electrodes that stimulate 4 targets (ABVN only, ATN only, ABVN plus ATN, and Sham).

DETAILED DESCRIPTION:
The demand for chronic pain treatment has demonstrated an unprecedented increase over the last several decades, in part contributing to an unsustainable surge in opioid prescriptions. Countless patients were escalated to prolonged, high-dose opioid regimens over years of treatment. By 2014, 5.4% of US adults were estimated to use prescription opioids on a long-term basis. As the harms of opioid proliferation became increasingly clear, a dramatic paradigm shift occurred in which these drugs came to be seen as often more dangerous than beneficial for chronic pain. New clinical guidelines highlighted the risks of high-dose regimens as well as limited benefits, particularly insufficient analgesia, associated with long-term use. According to this new perspective, the preferred therapeutic modality for many patients is to significantly reduce, or even completely stop, using opioids.

Stimulation of the ABVN has demonstrated additional benefits for reducing the need for opioids for pain as well as lessening opioid withdrawal symptoms. Clinical trials of ABVN stimulation as an adjunctive treatment for pain have noted decreased intake of tramadol , remifentanil, morphine, as well as naproxen plus tramadol. A pioneering study of electrical stimulation at the cymba conchae in eight persons with opioid use disorder found significantly reduced withdrawal symptoms: first, decreases in anxiety, craving for opioids, chills, nausea; second, reduced bone and joint pain. Results in follow-up clinical trials bolstered the efficacy of ABVN stimulation for opioid withdrawal . More recently, an open-label trial of simultaneous ABVN and trigeminal stimulation found reduced withdrawal symptoms and decreased need for morphine maintenance in newborns with neonatal opioid withdrawal syndrome . This method of simultaneous vagal and trigeminal stimulation via the external ear is known as transcutaneous auricular neurostimulation (tAN), as the targets of electrical stimulation include the ABVN and auriculotemporal nerve (ATN), which is a branch of the mandibular division of the trigeminal nerve. Electrodes applied to select dermatome regions can target ear neural structures and deliver non-invasive vagus nerve stimulation (VNS) and trigeminal nerve stimulation (TNS). See Figure 1.

Use of tAN devices for pain relief is an attractive alternative to pharmacologic and opioid-based approaches because it is safe and effective and presents no addiction liability. In order to increase clinical adoption and optimize efficacy of these devices, the mechanism of action must be fully characterized.

This study is investigating the mechanism behind tAN in a healthy cohort. Using tAN combined with advanced neuroimaging, we hope to begin to understand what parts of the brain are activated during tAN, compared to sham.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have the capacity and ability to provide one's own consent and sign the informed consent document

Exclusion Criteria:

* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
BOLD signal changes during stimulation relative to no stimulation | During tAN
  . tAN will will be administered to participants within the bore of the MRI scanner while we acquire high resolution functional neuroimaging. Both a general linear model and SNM approach will be used to examine BOLD signal changes during stimulation relative to rest blocks, comparing each of the four stimulation targets within- and between subjects to determine whether stimulating two cranial nerves produces a more robust neurophysiological effect than either single nerve or sham stimulation alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No